CLINICAL TRIAL: NCT04498754
Title: An Evaluation of Insomnia Treatment to Reduce Cardiovascular Risk in Patients With Posttraumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00100446
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Posttraumatic Stress Disorder; Cardiovascular Risk Factor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants who are originally assigned to the minimal contact control condition will be invited to receive the active condition treatment after their study involvement has been completed, but no additional data will be collected from them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy for Insomnia (CBT-I) (Experimental): Participants assigned to this arm will receive eight sessions of a well-established, evidence-based therapy called cognitive behavior therapy for insomnia (CBT-I).
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia
- Minimal Contact Control Condition (Other): Participants assigned to this condition will be contacted every week for eight weeks and monitored regarding their insomnia symptoms.
  Interventions: Behavioral: Weekly phone contacts

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Insomnia — 8 sessions of treatment for insomnia.
  Other Names: CBT-I
  Arms: Cognitive Behavior Therapy for Insomnia (CBT-I)
Behavioral: Weekly phone contacts — Weekly calls to monitor insomnia symptoms.
  Arms: Minimal Contact Control Condition

SUMMARY:
Posttraumatic stress disorder (PTSD) is a chronic, debilitating psychiatric disorder that is associated with an increased risk of death due to cardiovascular disease (CVD). Most individuals with PTSD also have Insomnia Disorder. Sleep quality is also associated with risk factors for CVD. The objective of this study is to examine how insomnia contributes to CVD risk among people with PTSD. The investigators will also examine whether this risk can be decreased with treatment for Insomnia Disorder.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a disabling and costly psychiatric disorder that is estimated to occur in 20% of individuals who are exposed to a traumatic event and is chronic in one third of cases. In addition to its negative impact on quality of life, there is substantial evidence that PTSD (even after controlling for depression and other risk factors) is associated with a markedly increased risk of cardiovascular morbidity and mortality. However, the mechanisms for the association between PTSD and cardiovascular disease (CVD) risk are not well understood. Although adverse health behaviors, including cigarette smoking, alcohol abuse and poor medication adherence are common in PTSD, recent prospective studies show that they do not account for the magnitude of CVD risk among individuals with PTSD. The investigators propose to test our central hypothesis by evaluating whether CBT-I results in improved biomarkers of CVD risk among those with PTSD. Well established biomarkers of CVD related morbidity and mortality will be used including measures of vascular endothelial function measured by brachial artery flow-mediated dilation (FMD), nighttime blood pressure (BP) dipping measured using 24-hour ambulatory blood pressure monitoring (ABPM), and sympathetic nervous system (SNS) activity as measured by 24-hour urinary catecholamines. Investigators will also assess lipid profile, which along with BP is a modifiable component with marked impact on the atherosclerotic cardiovascular disease (ASCVD) risk score. The primary sleep parameter of interest is objectively-measured sleep efficiency (through actigraphy), although self-report insomnia measures and sleep related arousal will also be measured. The rationale for the proposed research is that once it is established that insomnia is an important and modifiable symptom conveying increased CVD risk in this population, the development of new and innovative approaches to integrating insomnia treatment with PTSD-focused interventions can be developed. 150 men and women with comorbid PTSD and insomnia disorder will be randomly assigned with a 2:1 ratio to 8-week cognitive behavioral therapy-Insomnia (CBT-I) intervention or a waiting period control condition. Sleep quality parameters and CVD risk biomarkers will be assessed at pre-randomization baseline, post-intervention, and at a 6-month follow-up. The study is designed to evaluate the association between insomnia and CVD risk biomarkers among persons with PTSD, and determine whether improvements in insomnia symptoms are associated with improvements in CVD risk biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Is between 40-59 years old;
* Has a current diagnosis of chronic PTSD (at least 3 months duration) based on the Clinician Administered PTSD Scale DSM-5 version (Weathers et al., 2013);
* Has a current diagnosis of ID as defined in the International Classification of Sleep Disorders (ICSD-3; American Academy of Sleep Medicine, 2014)

Exclusion Criteria:

* Has a history of CVD events, including myocardial infarction, stroke, transient ischemic attack, or coronary revascularization;
* Has diagnosis of congestive heart failure or coronary artery disease based on results of diagnostic testing;
* Has a current alcohol use or substance use disorder (those who meet lifetime but not current alcohol or substance use disorder will be included);
* Is currently participating in or has recently (past 6 months) participated in an evidence-based trauma focused therapy for PTSD;
* Has cognitive impairment as evidenced by less than 20 on the Montreal Cognitive Assessment scale (M0CA; Nasreddine et al., 2005);
* Meets criteria for a psychotic spectrum disorder or bipolar disorder;
* Has severely impaired hearing or speech;
* Is pregnant;
* Does not use benzodiazepines for sleep, and if prescribed benzodiazepines for some other use (e.g., anxiety, panic attacks), uses them fewer than four times in a one month period.;
* Is not stable (medications and dose stable for one month) on any other current psychoactive and/or cardiovascular medications or will not be stable on these medications during the course of the study;
* Works night shift;
* Is participating in another interventional study to address insomnia;
* Has prominent suicidal or homicidal ideation (as assessed through a clinical interview);
* Has a serious/terminal illness or other health problem that would prohibit participation in the study;
* Has nonclinically significant or sub-threshold insomnia as indicated by a score of <8 on the Insomnia Severity Index;
* Has seizures (based on clinical interview and self-report);
* Has a body mass index of 45 or greater;
* Has sleep apnea (based on the overnight assessment described below) or a positive sleep apnea screen;
* Has restless leg syndrome (based on the Duke Structured Interview for Sleep Disorders (DSISD); Edinger, Wyatt, & Olsen, 2009), and that sleep disorder is the primary cause of their sleep complaint (participants with restless legs syndrome who also have insomnia disorder can be included in the study);
* Has an organic cause of sleep disruption that cannot be addressed by cognitive-behavioral changes (e.g., hyperthyroidism), as determined by the DSISD;
* Has excessive daytime sleepiness, defined as a score >15 on the Epworth Sleepiness Scale (ESS) or as determined by the DSISD;
* Does not complete sleep diary assessments within 6 hours of rising on at least 5 of the 7 days of the initial assessment period; or
* Cancels or no-shows for two or more Time 1 assessment appointments
* Has uncontrolled hypertension (screening office BP > 160/100 mm Hg)

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in nighttime blood pressure | Baseline and post-treatment (approximately eight weeks)
  Nighttime systolic and diastolic blood pressure measured by 24-hour ambulatory blood pressure monitor.
Change in nighttime blood pressure | Baseline and 6-month follow-up
  Nighttime systolic and diastolic blood pressure measured by 24-hour ambulatory blood pressure monitor.
Change in nighttime blood pressure dipping | Baseline and post-treatment (approximately eight weeks)
  Systolic and diastolic blood pressure dipping measured by 24-hour ambulatory blood pressure monitoring, and defined as the percent change in blood pressure from the wake period to the nighttime sleep period.
Change in nighttime blood pressure dipping | Baseline and 6-month follow-up
  Systolic and diastolic blood pressure dipping measured by 24-hour ambulatory blood pressure monitoring, and defined as the percent change in blood pressure from the wake period to the nighttime sleep period.
Change in vascular endothelial function | Baseline and post-treatment (approximately eight weeks)
  Vascular endothelial function will be measured by vascular ultrasound to determine flow mediated dilation (FMD) of the brachial artery. V
Change in vascular endothelial function | Baseline and 6-month follow-up
  Vascular endothelial function will be measured by vascular ultrasound to determine flow mediated dilation (FMD) of the brachial artery.
Change in nighttime sympathetic nervous system activity | Baseline and post-treatment (approximately eight weeks)
  Measured by 24 hour urine collection (awake and sleep period collection separated) assayed for catecholamines (epinephrine, norepinephrine) and creatinine.
Change in nighttime sympathetic nervous system activity | Baseline and 6-month follow-up
  Measured by 24 hour urine collection (awake and sleep period collection separated) assayed for catecholamines (epinephrine, norepinephrine) and creatinine.
Change in 10-year atherosclerotic cardiovascular disease risk | Baseline and post-treatment (approximately eight weeks)
  The risk of having a primary atherosclerotic cardiovascular disease event within 10 years will be based upon the pooled cohort equations model developed by the American College of Cardiology/American Heart Association.
Change in 10-year atherosclerotic cardiovascular disease risk | Baseline and 6-month follow-up
  The risk of having a primary atherosclerotic cardiovascular disease event within 10 years will be based upon the pooled cohort equations model developed by the American College of Cardiology/American Heart Association.
Change in insomnia severity | Baseline and post-treatment (approximately eight weeks)
  Insomnia measured by the Insomnia Severity Index. The measure has a score range from 0 to 28, with higher scores indicating more severe insomnia.
Change in insomnia severity | Baseline and 6-month follow-up
  Insomnia measured by the Insomnia Severity Index. The measure has a score range from 0 to 28, with higher scores indicating more severe insomnia.
Change in sleep efficiency | Baseline and post-treatment (approximately eight weeks)
  Sleep efficiency (percent-time asleep during the sleep period) measured by sleep diary and wrist actigraphy.
Change in sleep efficiency | Baseline and 6-month follow-up
  Sleep efficiency (percent-time asleep during the sleep period) measured by sleep diary and wrist actigraphy.

SECONDARY OUTCOMES:
Change in subjective sleep quality | Baseline and 6-month follow-up
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index. The scale has a score range of 0 to 21, with lower scores on this measure indicating better sleep quality.
Change in subjective sleep quality | Baseline and post-treatment (approximately eight weeks)
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index.scale has a score range of 0 to 21, with lower scores on this measure indicating better sleep quality.
Change in quality of life | Baseline and 6-month follow-up
  Quality of life will be measured using the Short Form-36 Health Survey. Scores on this measure range from 0 to 100, with higher scores indicating better quality of life.
Change in quality of life | Baseline and post-treatment (approximately eight weeks)
  Quality of life will be measured using the Short Form-36 Health Survey. Scores on this measure range from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Beckham, PhD, Principal Investigator — Duke Health; Andrew Sherwood, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04498754/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04498754/ICF_001.pdf